CLINICAL TRIAL: NCT01993498
Title: A Prospective Cohort to Investigate Survivorship Issues in Patients With Early Cancer
Brief Title: Chronic Toxicities Related to Treatment in Patients With Localized Cancer
Acronym: CANTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UC-0140/1103 CANTO; 2011-A01095-36 (Other: French Conpetant Authority)
Record Dates: First submitted 2013-10-17; First posted 2013-11-25 (Estimated); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Nos Metastatic Recurrent; Early Lung Cancer
Keywords: cancer toxicities; cohort; breast cancer; early lung cancer
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: For each patient, in addition to standard medical follow-up collected at selection, and yearly after acute treatment cancer phase during 5 years, the CANTO-specific follow-up includes 16 patient-reported questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- breast cancer treatment + blood sampling (Other): Standard treatment of breast cancer with intervention : samples collection
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — blood samples collection

SUMMARY:
The aims of the cohort will be to quantify impact of cancer treatments toxicities , and to generate predictors of chronic toxicity in patients with non-metastatic cancer. Study of the original cohort will be focused on localized breast cancer patients, other localisation in non-metastatic setting will be explored furtherwise, fist of all in lung cancer.

The project will include four specific aims :

1. To develop a database of chronic treatment related toxicity in a cohort of 14750 women with stage I-III breast cancer (= non metastatic), whatever these treatments are (surgery; radiation therapy; chemotherapy …)
2. To describe incidence, clinical presentation, and outcome of chronic toxicities.
3. To describe the psychological, the social and the economic impacts of chronic toxicities.
4. To generate predictors for chronic toxicities in order to prevent them, based upon biological criteria.

The expected impact of these toxicities, when identified, will be to improve quality of life and to decrease health cost, by the early identification of patients at high risk of toxicity. Such early identification could lead to prevent toxic effect by: a. developing prevention strategies, b. substituting toxic treatment by a non (less) toxic one.

Also, such cohort will offer a quantification of the impact of treatment toxicity, that could be further used to quantify medical usefulness of strategies that aim at decreasing treatment toxicities (implementation of predictive biomarker for resistance, cytotoxic-free regimen etc…)

DETAILED DESCRIPTION:
SPECIFIC AIM I: TO DEVELOP A TOXICITY DATABASE ON A COHORT OF 20,000 WOMEN WITH STAGE I-III (NON METASTATIC) BREAST CANCER

Selection criteria The cohort will include female patients with non-metastatic breast cancer (stage I-III) without any selection based on their characteristics (except stage) or treatment. They may be included in other concomitant clinical studies.

Patients will have to sign informed consent and will have to benefit from social security.

The lack of selection criteria is related to the fact that the cohort aims at investigating toxicity in the whole population of breast cancer from a public health perspective.

Sample size The cohort plans to include 14750 women in 13 years. A cohort of 14750 patients will allow to detect a two fold increased in the risk of a specific toxicity in a homogenous subgroup.

As illustration, the study present a 90% power to detect whether a variable (age as example) observed in 50% of patients is associated with an increased risk of toxicity (heart toxicity) in a specific subgroup (Her2+++).

Development of the cohort The14750 patients will be recruited in 26 cancer centers, maximum in France. These patients will be followed for at least 5 years in the context of the cohort. After 5 years, additional specific data will then be captured each year.

Patients will be included at the time of diagnosis, before any cancer specific treatment. After having signed informed consent, the patient will fill a first questionnaire for demographics (adapted from French DREES reference study) and living conditions, and a set of validated questionnaires related to QoL and special psychological dimensions. In addition, blood samples will be collected at baseline.

The toxicities (events) will start to be collected 3 months after the end of "acute" treatment (surgery/adjuvant/chemotherapy/radiation therapy). Toxicity data will also be collected at the time of the last chemotherapy. Toxicities will be collected each 6 months, alternatively by a dedicated nurse and by the patient herself. Three sets of toxicities will be collected.

* First, predefined and previously described toxicities will be collected on dedicated items in the case report form.
* Second, unknown toxicities will be captured by the use of a patient's notebook where each patient will collect events and doctor' visits (general practitioner or organ specialist). This will allow capturing events that have not previously been associated with cancer treatment toxicities.
* Finally, objective measurements by paraclinic exams will be done. This includes yearly blood tests and a heart ultrasonography at 1 and 5 years.

In addition to the data collection, a baseline blood sample for genetic analyses will be done, and serum samples will be collected at baseline and yearly during 5 years (serum).

Outcome data will also be collected and will include metastatic relapse (+ site), locoregional relapse (+ site) and death.

SPECIFIC AIM II: TO DESCRIBE INCIDENCE, CLINICAL PRESENTATION, BIOLOGICAL CHARACTERISTICS AND OUTCOME OF CHRONIC TOXIC EVENTS

This specific aim will follow three goals :

* First, the investigators will describe the incidence of predefined chronic toxicities according to the treatment received.
* Second, the investigators will aim at identifying new treatment-related toxicities. This information will be captured through a dedicated notebook where each patient will report all health and social related events.
* Finally, the investigators will also assess the outcome of each adverse event, and try to develop some hypotheses to be addressed in further clinical trials.

SPECIFIC AIM III: TO DESCRIBE THE PSYCHOLOGICAL AND THE SOCIAL IMPACTS OF TOXIC EVENTS This specific aim will be split in two parts: a. to describe the psychological and the social impact to the patient, b. to describe the impact at the population level.

To describe psychological and social impact for the patient

Using robust well validated methods, subjective and objective dimensions of wellbeing will be investigated, that is: a. Quality of life b. Living conditions c. Psychosocial issues.

Quality of life Global perception of quality of life will be assessed through different survey

Social impact Living conditions will be assessed through a questionnaire derived from the French DRESS reference study on living conditions. The initial questionnaire was designed by DRESS to investigate the social, economical, professional condition two years after the diagnosis of cancer: back or abandonment of the initial professional/social activity, conversion, income trends, etc.

Psychological impact This part will focus on psychological functioning, including psychological impact of chronic toxicities and psychological impact of cancer itself. Psychological impact is mainly expected on emotional issues, cognitive disorders, body image and sexual disorders.

To describe the impact on the society This sub-aim will mainly focus on medico-economics and will assess the global impact of treatment toxicity on health economy. The quantification of costs related to toxicities is a major challenge since it could allow to identify avoidable major source of expenses and could allow better tailoring treatment accordingly. Specific partnerships are being developed with the French social security and other public/private partners in order to accurately quantify toxicity-related cost.

SPECIFIC AIM IV TO DEVELOP PREDICTORS FOR CHRONIC TOXICITIES In the present specific aim, the goal will be to develop molecular/biologic predictors for toxic events. In as many cases as possible, the investigators will split the cohort into a discovery set and a test set, or will identify a cross-validating series before doing analyses.

Ultimately, the goal is to develop multiparametric scores to predict the occurrence of toxicity.

Regarding molecular predictors, it is planned that 20 ml blood will be collected yearly. One sample at baseline will be dedicated to single nucleotide polymorphism (SNP) arrays and validation of candidate genetic variants.

A number of tests are already planned. First, we will investigate conventional biological parameters including endocrine tests (cortisolemia, TSH, estradiol levels, mullerian hormone…), metabolic test (including lipidemia), hematologic tests, liver function, immune function (assessed by lymphocyte counts). Second, more recent and under investigation tests will be added including troponin (heart failure), mullerian hormone, bone resorption markers (bone loss), RANK / RANKL, osteoprotegerin (bone loss).

Finally, it is planned to use the baseline sample for the discovery of genetic tests and to use the serum for the discovery of biochemical predictors.

ELIGIBILITY:
CANTO - Breast

Inclusion Criteria:

* Women,
* Aged 18 years and over,
* With an invasive breast cancer diagnosed by cytology or histology,
* No clinical evidence of metastasis at the time of inclusion,
* Untreated including scored for breast cancer surgery in progress,
* Patient receiving a social security system,
* Patient mastering the French language,
* Free and informed consent for additional biological samples, different questionnaires and collecting information on resource usage.
* (Since february 2022) Patient :

  1. Age < 45 years at diagnostic
  2. Or CT2-3, cN0-3, HER2+(RH+or RH-) or RH-HER2-
  3. Or Eligible to Pembrozilumab, Olaparib, TDM1, Abemaciclib or Ribociclib

Exclusion Criteria:

* Metastatic breast cancer,
* Local recurrence of breast cancer,
* History of cancer within 5 years prior to entry into the trial other than basal cell skin or carcinoma in situ of the cervix,
* Already received treatment for breast cancer ongoing,
* Blood transfusion performed for less than six months,
* Persons deprived of liberty or under supervision (including guardianship).

CANTO - Lung

Inclusion Criteria:

* Aged 18 years and over, Having lung cancer diagnosed by cytology or histology or suspected cancer of the lung,
* Tumor cTX to cT4, cN0-3,
* No clinical evidence of metastasis at the time of inclusion (patients with metastases on extension assessment within 6 months following diagnosis will be removed from the study),
* Eligible for curative treatment by surgery or radiotherapy * (note patients treated with exclusive chemotherapy, exclusive radiotherapy or exclusive stereotactic radiotherapy will be out of study)
* Lack of treatment received for current lung cancer, including surgical treatment
* Patient benefiting from a social protection scheme,
* Patient mastering the French language,
* Free and informed consent for additional biological samples, the different questionnaires and the collection of information on resource consumption.

Exclusion Criteria:

* Metastatic lung cancer,
* Local relapse of lung cancer,
* History of cancer within 3 years prior to study entry other than basal cell cutaneous or epithelioma in situ of the cervix,
* Treatment already received for current lung cancer,
* Blood transfusion carried out less than 6 months ago,
* Persons deprived of liberty or under guardianship (including curatorship).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14750 (Estimated)
Dates: Start 2012-02-20 (Actual); Primary Completion 2034-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of chronic toxicity in patients treated for non-metastatic breast cancer | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Inès VAZ-LUIS, Professor, Study Director — Gustave Roussy - Villejuif
Locations (1):
- Gustave roussy, Villejuif, France

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.

REFERENCES:
- [Derived] Bidard FC, Gessain G, Bachelot T, Frechin L, Vincent-Salomon A, Drubay D, Lemonnier J, Walter T, Penault-Llorca F, Martin AL, Gaudin C, Bichat A, Sassi F, Berlemont S, Chavez-MacGregor M, Rugo HS, Badoual C, Pistilli B, Ribeiro J, Di Meglio A, Lacroix-Triki M, Vaz Luis I, Lerousseau M, Andre F. Identifying Patients With Low Relapse Rate Despite High-Risk Estrogen Receptor-Positive/Human Epidermal Growth Factor Receptor 2-Negative Early Breast Cancer: Development and Validation of a Clinicopathologic Assay. J Clin Oncol. 2025 Oct;43(28):3090-3101. doi: 10.1200/JCO-25-00742. Epub 2025 Aug 22. PMID 40845255
- [Derived] Giugliano F, Bertaut A, Blanc J, Martin AL, Gaudin C, Fournier M, Kieffer A, Sauterey B, Levy C, Campone M, Tarpin C, Lerebours F, Mouret-Reynier MA, Curigliano G, Andre F, Pistilli B, Rassy E. Characteristics, treatment patterns and survival of patients with high-risk early hormone receptor-positive breast cancer in French real-world settings: an exploratory study of the CANTO cohort. ESMO Open. 2024 Dec;9(12):103994. doi: 10.1016/j.esmoop.2024.103994. Epub 2024 Nov 28. PMID 39612621
- [Derived] Pagliuca M, Havas J, Thomas E, Drouet Y, Soldato D, Franzoi MA, Ribeiro J, Chiodi CK, Gillanders E, Pistilli B, Menvielle G, Joly F, Lerebours F, Rigal O, Petit T, Giacchetti S, Dalenc F, Wassermann J, Arsene O, Martin AL, Everhard S, Tredan O, Boyault S, De Laurentiis M, Viari A, Deleuze JF, Bertaut A, Andre F, Vaz-Luis I, Di Meglio A. Long-term behavioral symptom clusters among survivors of early-stage breast cancer: Development and validation of a predictive model. J Natl Cancer Inst. 2025 Jan 1;117(1):89-102. doi: 10.1093/jnci/djae222. PMID 39250750
- [Derived] Sandoval JL, Franzoi MA, di Meglio A, Ferreira AR, Viansone A, Andre F, Martin AL, Everhard S, Jouannaud C, Fournier M, Rouanet P, Vanlemmens L, Dhaini-Merimeche A, Sauterey B, Cottu P, Levy C, Stringhini S, Guessous I, Vaz-Luis I, Menvielle G. Magnitude and Temporal Variations of Socioeconomic Inequalities in the Quality of Life After Early Breast Cancer: Results From the Multicentric French CANTO Cohort. J Clin Oncol. 2024 Aug 20;42(24):2908-2917. doi: 10.1200/JCO.23.02099. Epub 2024 Jun 18. PMID 38889372
- [Derived] Balazard F, Bertaut A, Bordet E, Mulard S, Blanc J, Briot N, Paux G, Dhaini Merimeche A, Rigal O, Coutant C, Fournier M, Jouannaud C, Soulie P, Lerebours F, Cottu PH, Tredan O, Vanlemmens L, Levy C, Mouret-Reynier MA, Campone M, Brady KJS, Sasane M, Rice M, Coulouvrat C, Martin AL, Jacquet A, Vaz-Luis I, Herold C, Pistilli B. Adjuvant endocrine therapy uptake, toxicity, quality of life, and prediction of early discontinuation. J Natl Cancer Inst. 2023 Sep 7;115(9):1099-1108. doi: 10.1093/jnci/djad109. PMID 37434306
- [Derived] Ghannam Y, Di Meglio A, Sarrade T, Jacquet A, Everhard S, Kirova Y, Peignaux K, Guilbert P, Charra-Brunaud C, Blanchecotte J, Bochaton OF, Pasquier D, Racadot S, Bourgier C, Geffrelot J, Benyoucef A, Paris F, Auzac G, Luis IV, Rivera S. Impact of radiation therapy on fatigue at 1 year in breast cancer survivors in the prospective multicentre CANcer TOxicity cohort. Eur J Cancer. 2022 Dec;177:143-153. doi: 10.1016/j.ejca.2022.09.026. Epub 2022 Oct 10. PMID 36356418
- [Derived] Soldato D, Havas J, Crane TE, Presti D, Lapidari P, Rassy N, Pistilli B, Martin E, Del Mastro L, Martin AL, Jacquet A, Coutant C, Cottu P, Merimeche A, Lerebours F, Tredan O, Vanlemmens L, Andre F, Vaz-Luis I, Di Meglio A. Coffee and tea consumption, patient-reported, and clinical outcomes in a longitudinal study of patients with breast cancer. Cancer. 2022 Oct 1;128(19):3552-3563. doi: 10.1002/cncr.34401. Epub 2022 Aug 1. PMID 35913436
- [Derived] Presti D, Havas J, Soldato D, Lapidari P, Martin E, Pistilli B, Jouannaud C, Emile G, Rigal O, Fournier M, Soulie P, Mouret-Reynier MA, Tarpin C, Campone M, Guillermet S, Martin AL, Everhard S, Di Meglio A. Factors associated with enrolment in clinical trials among women with early-stage breast cancer. ESMO Open. 2022 Jun;7(3):100513. doi: 10.1016/j.esmoop.2022.100513. Epub 2022 Jun 17. PMID 35724624
- [Derived] Baker JL, Di Meglio A, Gbenou AS, El Mouhebb M, Iyengar NM, Michiels S, Cottu P, Lerebours F, Coutant C, Lesur A, Tredan O, Vanlemmens L, Jouannaud C, Hrab I, Everhard S, Martin AL, Arveux P, Fabrice A, Vaz-Luis I, Jones LW. Association between physical activity and neoadjuvant chemotherapy completion and pathologic complete response in primary breast cancer: the CANTO study. Br J Cancer. 2022 Sep;127(5):886-891. doi: 10.1038/s41416-022-01870-y. Epub 2022 Jun 17. PMID 35715631
- [Derived] Di Meglio A, Havas J, Gbenou AS, Martin E, El-Mouhebb M, Pistilli B, Menvielle G, Dumas A, Everhard S, Martin AL, Cottu PH, Lerebours F, Coutant C, Lesur A, Tredan O, Soulie P, Vanlemmens L, Joly F, Delaloge S, Ganz PA, Andre F, Partridge AH, Jones LW, Michiels S, Vaz-Luis I. Dynamics of Long-Term Patient-Reported Quality of Life and Health Behaviors After Adjuvant Breast Cancer Chemotherapy. J Clin Oncol. 2022 Sep 20;40(27):3190-3204. doi: 10.1200/JCO.21.00277. Epub 2022 Apr 21. PMID 35446677
- [Derived] Vaz-Luis I, Di Meglio A, Havas J, El-Mouhebb M, Lapidari P, Presti D, Soldato D, Pistilli B, Dumas A, Menvielle G, Charles C, Everhard S, Martin AL, Cottu PH, Lerebours F, Coutant C, Dauchy S, Delaloge S, Lin NU, Ganz PA, Partridge AH, Andre F, Michiels S. Long-Term Longitudinal Patterns of Patient-Reported Fatigue After Breast Cancer: A Group-Based Trajectory Analysis. J Clin Oncol. 2022 Jul 1;40(19):2148-2162. doi: 10.1200/JCO.21.01958. Epub 2022 Mar 15. PMID 35290073
- [Derived] Di Meglio A, Charles C, Martin E, Havas J, Gbenou A, Flaysakier JD, Martin AL, Everhard S, Laas E, Chopin N, Vanlemmens L, Jouannaud C, Levy C, Rigal O, Fournier M, Soulie P, Scotte F, Pistilli B, Dumas A, Menvielle G, Andre F, Michiels S, Dauchy S, Vaz-Luis I. Uptake of Recommendations for Posttreatment Cancer-Related Fatigue Among Breast Cancer Survivors. J Natl Compr Canc Netw. 2022 Feb 7;20(13). doi: 10.6004/jnccn.2021.7051. PMID 35130491
- [Derived] Di Meglio A, Havas J, Soldato D, Presti D, Martin E, Pistilli B, Menvielle G, Dumas A, Charles C, Everhard S, Martin AL, Coutant C, Tarpin C, Vanlemmens L, Levy C, Rigal O, Delaloge S, Lin NU, Ganz PA, Partridge AH, Andre F, Michiels S, Vaz-Luis I. Development and Validation of a Predictive Model of Severe Fatigue After Breast Cancer Diagnosis: Toward a Personalized Framework in Survivorship Care. J Clin Oncol. 2022 Apr 1;40(10):1111-1123. doi: 10.1200/JCO.21.01252. Epub 2022 Jan 21. PMID 35061509
- [Derived] Caumette E, Vaz-Luis I, Pinto S, Havas J, Bovagnet T, Ruiz de Azua G, Di Meglio A, Martin AL, Everhard S, Cottu P, Vanlemmens L, Jouannaud C, Lerebours F, Dumas A, Menvielle G. The Challenge of Return to Work after Breast Cancer: The Role of Family Situation, CANTO Cohort. Curr Oncol. 2021 Oct 1;28(5):3866-3875. doi: 10.3390/curroncol28050330. PMID 34677248
- [Derived] Di Meglio A, Gbenou AS, Martin E, Pistilli B, Ligibel JA, Crane TE, Flaysakier JD, Minvielle E, Vanlemmens L, Guenancia C, Rigal O, Fournier M, Soulie P, Mouret-Reynier MA, Tarpin C, Boiffard F, Guillermet S, Everhard S, Martin AL, Giacchetti S, Petit T, Dalenc F, Rouanet P, Arnaud A, Andre F, Vaz-Luis I. Unhealthy behaviors after breast cancer: Capitalizing on a teachable moment to promote lifestyle improvements. Cancer. 2021 Aug 1;127(15):2774-2787. doi: 10.1002/cncr.33565. Epub 2021 Apr 22. PMID 33887074
- [Derived] Di Meglio A, Menvielle G, Dumas A, Gbenou A, Pinto S, Bovagnet T, Martin E, Ferreira AR, Vanlemmens L, Arsene O, Ibrahim M, Wassermann J, Martin AL, Lemonnier J, Del Mastro L, Jones LW, Partridge AH, Ligibel JA, Andre F, Michiels S, Vaz Luis I. Body weight and return to work among survivors of early-stage breast cancer. ESMO Open. 2020 Nov;5(6):e000908. doi: 10.1136/esmoopen-2020-000908. PMID 33172957
- [Derived] Pistilli B, Paci A, Ferreira AR, Di Meglio A, Poinsignon V, Bardet A, Menvielle G, Dumas A, Pinto S, Dauchy S, Fasse L, Cottu PH, Lerebours F, Coutant C, Lesur A, Tredan O, Soulie P, Vanlemmens L, Jouannaud C, Levy C, Everhard S, Arveux P, Martin AL, Dima A, Lin NU, Partridge AH, Delaloge S, Michiels S, Andre F, Vaz-Luis I. Serum Detection of Nonadherence to Adjuvant Tamoxifen and Breast Cancer Recurrence Risk. J Clin Oncol. 2020 Aug 20;38(24):2762-2772. doi: 10.1200/JCO.19.01758. Epub 2020 Jun 22. PMID 32568632
- [Derived] Kabore EG, Guenancia C, Vaz-Luis I, Di Meglio A, Pistilli B, Coutant C, Cottu P, Lesur A, Petit T, Dalenc F, Rouanet P, Arnaud A, Arsene O, Ibrahim M, Wassermann J, Boileau-Jolimoy G, Martin AL, Lemonnier J, Andre F, Arveux P. Association of body mass index and cardiotoxicity related to anthracyclines and trastuzumab in early breast cancer: French CANTO cohort study. PLoS Med. 2019 Dec 23;16(12):e1002989. doi: 10.1371/journal.pmed.1002989. eCollection 2019 Dec. PMID 31869400
- [Derived] Ferreira AR, Di Meglio A, Pistilli B, Gbenou AS, El-Mouhebb M, Dauchy S, Charles C, Joly F, Everhard S, Lambertini M, Coutant C, Cottu P, Lerebours F, Petit T, Dalenc F, Rouanet P, Arnaud A, Martin A, Berille J, Ganz PA, Partridge AH, Delaloge S, Michiels S, Andre F, Vaz-Luis I. Differential impact of endocrine therapy and chemotherapy on quality of life of breast cancer survivors: a prospective patient-reported outcomes analysis. Ann Oncol. 2019 Nov 1;30(11):1784-1795. doi: 10.1093/annonc/mdz298. PMID 31591636